CLINICAL TRIAL: NCT06068127
Title: Retrospective Study of Per-oral Endoscopic Pyloromyotomy (G-POEM) in Patients With Refractory Gastroparesis After Esophagectomy With Gastric Pull-through
Brief Title: G-POEM for Refractory Gastroparesis After Esophagectomy With Gastric Pull-through
Acronym: GESOM
Status: Recruiting | Type: Observational
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Doc. (Ass. prof.) Jan Martinek, MD, PhD, AGAF, Prof. Jan Martínek, MD, PhD, AGAF, Institute for Clinical and Experimental Medicine
Other Study IDs: GESOM
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Gastroparesis; Esophageal Cancer
MeSH Terms: conditions — Gastroparesis; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study assessing the effectiveness of endoscopic pyloromyotomy in patients suffering from gastroparesis and/or symptoms of delayed gastric emptying after esophagectomy with gastric pull-through. Several, mainly European, centres which perform G-POEM on a routine basis will be asked to participate. The main reason to assess the effectiveness of G-POEM in this specific subgroup of patients is the fact this specific subgroup of patients is often being excluded from trials assessing efficacy and safety of G-POEM.

The participating centres will be asked to report appropriate patients among those who have undergone G-POEM since 2015 till December 2023. Patients fulfilling inclusion and not having exclusion criteria will be included into the analysis; the minimum follow-up is set to 6 months after G-POEM. The main outcome is the symptomatic response at 6, 12 and 24 months (measured by GCSI score). Other endpoints will be change in other symptoms not covered by GCSI, change in gastric emptying rate and safety of the procedure.

For each enrolled patient a case report form (CRF) will be filled in and delivered to the leading centre via an online database or in other forms if preferred by the respective centres. The leading centre will be responsible for data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent G-POEM after esophagectomy with a gastric pull-through for confirmed (scintigraphy or breath test) or presumed gastroparesis. (Some centres perform G-POEM in patients whose gastroparesis was not confirmed by a scintigraphy or a breath test, therefore it is only presumed. This particular subset of patients will be analysed separately.)
* Total GCSI score before G-POEM at least 1.0.
* At least 6 months follow-up after G-POEM.

Exclusion Criteria:

* Organic pyloric obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent G-POEM after esophagectomy with a gastric pull-through in any of the participating centers since January 2015 till December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2024-03-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
GCSI score | At baseline and 3, 6, 12, 24, 36 months after G-POEM
  Gastroparesis Cardinal Symptom Index questionnaire: The score ranges from 0 to 5 for each symptom (9 questions) and these are averaged into subscores and into a total score (also ranging from 0 to 5). Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Gastric emptying by scintigraphy | At baseline and 3, 6, 12, 24, 36 months after G-POEM
  Gastric scintigraphy protocol endorsed by both American Neurogastroenterology and Motility Society and American Nuclear Medicine Society will be used to assess gastric emptying with a standard 200 kcal, 2% fat egg-substitute test meal. Gamma camera images will be obtained immediately after meal ingestion and then at 1, 2, 3 and 4 hours. Diagnostic criterion for delayed gastric emptying is defined as the percentage of gastric retention >60% at 2 h or ≥ 10% at 4 h or both. Half-time (T1/2) emptying time will also be calculated. At least 72 hours before gastric emptying test, narcotics and other medications that can interfere with gastric emptying will be discontinued.
Gastric emptying by breath test | At baseline and 3, 6, 12, 24, 36 months after G-POEM
  Gastric emptying assessed using 13C breath test with octanoic acid. This measurement is an alternative to the measurement of gastric emptying by scintigraphy. The choice depends on the practice in a particular center.
Pyloric distensibility | At baseline and 3, 6, 12, 24, 36 months after G-POEM
  Pyloric distensibility measured by impedance planimetry (EndoFLIP device)

CONTACTS AND LOCATIONS:
Locations (2):
- Institute for Clinical and Experimental Medicine, Prague, Czechia
- Hôpital Nord, Marseille, France